CLINICAL TRIAL: NCT05467579
Title: Short-term and Long-term Evaluation of Three-dimensional Morphological Condylar and Mandibular Changes in Patients Affected by Juvenile Idiopathic Arthritis Treated With Mandibular Advancement Clear Aligner. A Prospective Controlled Study
Brief Title: Mandibular Advancement Clear Aligner Treatment in Juvenile Idiopathic Arthritis Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Genova (Other)
Collaborators: University of Milan - Prof. Maspero Cinzia (Unknown); University of Milan - Dr. Abate Andrea (Unknown)
Responsible Party: Principal Investigator, ALESSANDRO UGOLINI, Professor, University of Genova
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 072022
Record Dates: First submitted 2022-07-14; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Juvenile Idiopathic Arthritis; Malocclusion, Angle Class II
MeSH Terms: conditions — Arthritis, Juvenile; Malocclusion, Angle Class II | interventions — Activator Appliances

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Active Comparator): Healthy patients that will serve as controls will recruited having the same demographic characteristics of the experimental group i.e., age, sex, vertebral maturation stage and the same cranio-facial features, skeletal class II, class II division 1 malocclusion, mandibular retrognathia, normal/hyperdivergent growth pattern.
  Interventions: Device: Device: orthodontic - mandibular advancement clear aligner
- JIA subjects (Experimental): Young people aged from 10 to 14 years old with skeletal class II, class II division 1 malocclusion, mandibular retrognathia, normal/hyperdivergent growth pattern, and affected by juvenile idiopathic arthritis
  Interventions: Device: Device: orthodontic - mandibular advancement clear aligner

INTERVENTIONS:
Device: Device: orthodontic - mandibular advancement clear aligner — Intervention orthodontic - mandibular advancement: mandibular retrognathia correction with a mandibular advancement using a step-wise approach with clear aligner.
  Other Names: MA clear aligner; activator appliances

SUMMARY:
There is currently no information on how mandibular advancement therapy could influence three-dimensionally the condylar and mandibular morphology in growing patients affected by Juvenile Idiopathic Arthritis (JIA). Therefore, the aim is to assess the three-dimensional morphological mandibular changes produced by the Invisalign® Mandibular Advancement (MA) (Align Technology, San José, CA, USA) in growing subjects affected by juvenile idiopathic arthritis with unilateral and bilateral JIA and to compare them with not-JIA control subjects

DETAILED DESCRIPTION:
A wide range of functional appliances have been designed across the years to obtain a supplementary growth of the mandible by its forward posturing to correct mandibular retrusion. In a review published by Cozza et al., the efficiency of functional appliances used in healthy humans in terms of supplementary growth of the mandible per month of treatment, was measured. The Herbst appliance had the highest coefficient of efficiency (0.28 mm per month) followed by the Twin-block device (0.23 mm per month).

Different authors claimed that functional treatment by removable appliances may be effective in treating Class II malocclusion with clinically relevant skeletal effects if performed during the pubertal growth phase. However, the growth pattern in JIA patients is more complicated and difficult compared to the treatment groups in the above-mentioned studies. The pattern is not only characterized by a decrease in mandibular length, but also by a decreased ratio between the posterior and the anterior face height, due to a failure in the vertical growth of the condyles The favorable effect of functional orthopedic appliances in JIA cases is therefore, besides advancing the mandible, an anterior (counter clockwise) rotation with a possible increase of the posterior face height, if possible. The efficacy of the functional orthopedic appliance in the correction of open bite has been demonstrated by Ibitayo et al.

To date, different types of removable orthopedic appliances have been proposed into the scientific literature for management of deformities in skeletally immature patients with JIA, in particular the activator and the distraction splint. Although functional orthopedic treatment is recommended, literature is still lacking studies on this important topic.

Recently a mandibular advancement device (MA) was implemented by Align TechnologyTM (San José, CA, USA) on clear aligners, for the treatment of skeletal Class II in growing patients. Similarly, to the principle applied in Twin Block, MA is composed by two pairs of lateral inclined planes (precision wings), positioned buccally in the posterior area of aligners, which come into contact each time the patient closes his mouth determining a mandibular forward position.

Regarding the above-mentioned novel therapeutic approach, accurate bibliographic research performed on June 2022 showed that, the scientific literature needs further studies evaluating the skeletal effects produced by the Mandibular advancement with clear aligner since there is limited literature on its efficiency, consisting mostly of case studies. Recent longitudinal studies reported very promising results, when used in the pubertal growth phase. The short-term effects of Mandibular Advancement feature are dento-skeletal with additional growth of the mandible and improvement in facial convexity. The MA clear aligner treatment in JIA patients could bring countless benefits. The main ones are the possibility of performing a class II functional therapy with the same ability of a distraction splint or activators in promoting mandibular growth and at the same time controlling the vertical dimension with a programmed intrusion/extrusion of the teeth. Moreover, these therapeutic approaches should be more aesthetic, less bulky, and annoying appliances which can therefore guarantee greater collaboration from the patient. The latter would be reinforced by the fact that during functional therapy there would be a concomitant dental alignment with positive implications in patients whose facial aesthetics are already partially compromised, the face is one of the most salient and relevant social stimuli humans encounter and automatically evokes neural responses, facial deformity must not be underestimated. Moreover, clear aligner therapy is associated with minimal adverse events related to the periodontal structures compared to fixed appliances, this is of relevant interest in JIA subjects who often suffer from moderate or severe periodontitis.

ELIGIBILITY:
1. Aged from 10 to 14 years old and attending the Department of Biomedical Surgical and Dental Sciences, University of Milan at the peak of the pubertal spurt assessed using vertebral analysis.
2. Features of a class II, division 1 malocclusion with mandibular retrusion and ANB according to Riedel >4°.
3. Convex profile and minimum overjet of 4 mm in permanent dentition, without missing teeth
4. moderate crowding in the upper arch (≤4 mm)
5. Parental informed consent

Exclusion Criteria:

1. Previous orthodontic or orthopedic treatment with any type of intervention (to avoid confounding factors related to previous treatment)
2. Patients with severe transverse dental or skeletal discrepancies
3. Syndromes, orofacial cleft, or other special needs, except for Juvenile idiopathic arthritis
4. Missing teeth (to avoid confounding factors related to anchorage loss due to the absence or early extraction of permanent teeth)
5. Poor oral health that precludes orthodontic treatment (presence of caries, active white spots or periodontal diseases)

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of the facial profile | 12 months
  Clinical evaluation in vivo (binary outcome yes/no)
Mandibular growth achievement | 12 months
  Measured on CBCT scans (increase in mm of the mandibular length, superimposition of the 3D reconstruction of the condyles)
Presence of inflammation during active phase of mandibular advancement | 12 months
  To monitoring TMJ inflammation during the active phase of treatment comparing the MRI taken before the beginning of therapy with those taken as controls every six months until the end of treatment and to evaluate patient's reported outcomes regarding treatment with mandibular advancement both in JIA and in the healthy control group
Discomfort during active phase | 6 months
  Discomfort reported on a questionnaire during all the active phase of treatment recorded every 6 month (VAS scale, pain min-max 0-100)
Discomfort during active phase | 12 months
  Discomfort reported on a questionnaire during all the active phase of treatment recorded every 6 month (VAS scale, pain min-max 0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Milano, Ospedale maggiore Policlincio, IRCCS Cà Granda, Milan, Itali, Italy